CLINICAL TRIAL: NCT01007344
Title: A 4-week Study in Children and Adolescents With Familial or Severe Hypercholesterolemia Comparing Flaxseed Therapy to Placebo
Brief Title: Flaxseed Compared With Placebo in Patients With Hypercholesterolemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Brian McCrindle, Staff Cardiologist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1000008297
Record Dates: First submitted 2009-11-03; First posted 2009-11-04 (Estimated); Last update posted 2013-08-27 (Estimated); Status verified 2013-08

CONDITIONS: Familial or Severe Hypercholesterolemia
Keywords: flaxseed; hypercholesterolemia; children
MeSH Terms: conditions — Hypercholesterolemia | interventions — Linseed Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- flaxseed (Active Comparator): 2 muffins and 1 slice of bread for a total of 30g flaxseed per day
  Interventions: Dietary Supplement: flaxseed
- whole wheat flour (Placebo Comparator): 2 muffins and 1 slice of bread containing whole wheat flour per day
  Interventions: Dietary Supplement: whole wheat flour

INTERVENTIONS:
Dietary Supplement: flaxseed — 1 muffin for breakfast, 1 muffin for afternoon snack and 1 slice of bread for evening snack every day for 4 weeks
  Arms: flaxseed
Dietary Supplement: whole wheat flour — 1 muffin for breakfast, 1 muffin for afternoon snack and 1 slice of bread for evening snack every day for 4 weeks
  Arms: whole wheat flour

SUMMARY:
The aim of this study is to determine if thirty grams per day of flaxseed consumption for 4 weeks could potentially reduce the serum lipid levels in children and adolescents with familial or severe hypercholesterolemia compared to those on placebo.

DETAILED DESCRIPTION:
The proposed study is a 4 week randomized, double-blind, placebo-controlled clinical trial. Participants will be recruited from the pediatric lipid disorder clinic at the Hospital for Sick Children, which provides consultations to and management of children with primary lipid abnormalities. Patients that meet the study criteria will be approached during their routinely scheduled clinic visits, until the sample size (N=30) be reached. Patients will randomly be assigned to the intervention or the placebo group. The intervention group will be given muffins and breads containing ground flaxseed. Two muffins and one slice of bread will be consumed per day to provide a total of 30g flaxseed to the experimental group. The control group will be given muffins and breads containing whole wheat flour in place of flaxseed. Participants will be instructed to eat one muffin for breakfast, one muffin as an afternoon snack, and one slice of bread as an evening snack every day for a 4-week period. The muffins and breads use in the study will be baked by an independent baker.

ELIGIBILITY:
Inclusion Criteria:

* age 8 to 18 years
* positive first-degree family history of hypercholesterolemia or premature atherosclerotic cardiovascular disease
* elevated LDL level above 3.5 mmol/L and less than 5.0 mmol/L
* entered in the National Cholesterol Education Program Step II diet for at least 6 months

Exclusion Criteria:

* patients with secondary causes of hyperlipidemia
* history of major illness or surgery 3 months or less prior to enrollment
* taking lipid-lowering medications
* history of gastrointestinal problems
* allergies towards flaxseed

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2009-10; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
fasting serum total cholesterol, triglycerides, high-density lipoprotein (HDL) cholesterol, low-density lipoprotein (LDL) and C-reactive protein | 4 weeks

SECONDARY OUTCOMES:
LH (luteinizing hormone, FSH (follicle-stimulating hormone), DHEA-S (Dihydroepiandrosterone sulfate), free testosterone, androstenedione | 4 weeks
complete blood count | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Brian McCrindle, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Wong H, Chahal N, Manlhiot C, Niedra E, McCrindle BW. Flaxseed in pediatric hyperlipidemia: a placebo-controlled, blinded, randomized clinical trial of dietary flaxseed supplementation for children and adolescents with hypercholesterolemia. JAMA Pediatr. 2013 Aug 1;167(8):708-13. doi: 10.1001/jamapediatrics.2013.1442. PMID 23733031